CLINICAL TRIAL: NCT01418430
Title: HTLV-I Associated Adult T-cell Leukaemia/Lymphoma (ATLL) Pilot Study of Combination Therapy With CHOP-Zenapax (CHOP-daclizumab)
Brief Title: Pilot Study of Combination Therapy With CHOP-Zenapax (CHOP-daclizumab)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: King's College Hospital NHS Trust (Other)
Responsible Party: Dr Antonio Pagliuca, King's College Hospital NHS Foundation Trust
Purpose: Treatment
Other Study IDs: CHOP-Z
Record Dates: First submitted 2011-08-16; First posted 2011-08-17 (Estimated); Last update posted 2011-08-22 (Estimated); Status verified 2011-07

CONDITIONS: HTLV-I Associated Adult T-cell Leukaemia/Lymphoma (ATLL)
MeSH Terms: conditions — Lymphoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- CHOP-daclizumab (Experimental)
  Interventions: Drug: CHOP-daclizumab

INTERVENTIONS:
Drug: CHOP-daclizumab
  Other Names: CHOP-Zenapax

SUMMARY:
The purpose of this study is to determine the safety of the combination of CHOP plus daclizumab in patients with ATLL previously untreated with anthracycline based chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed ATLL requiring treatment

   1. Frank acute leukaemia or lymphoma subtypes
   2. Chronic and smouldering cases should be considered if they are symptomatic and require therapy, or there is evidence of disease progression
2. No previous treatment with anthracycline based cytotoxic chemotherapy

   a. Patients may have received interferon and /or zidovudine and/or non-anthracycline based therapy
3. Age 18-75 years
4. Written informed consent

Exclusion Criteria:

1. HIV 1 or 2 positivity
2. Pregnancy or breast-feeding
3. Concomitant chemo-radiotherapy
4. Prior hepatic or renal insufficiency with a bilirubin or transaminases greater than 5 times the normal range or a creatinine greater than 150μmol/l (not related to hypercalcaemia) following rehydration
5. Other concomitant neoplasms not related to HTLV-I
6. Cardiac or respiratory insufficiency with an ECOG score of greater than 3
7. Any serious active uncontrolled infection

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (1):
- King's College Hospital NHS Foundation Trust, London, United Kingdom